CLINICAL TRIAL: NCT03236025
Title: The Effectiveness of a Video-led Smoking Cessation Intervention in Helping Male Smokers in Mainland China Whose Partner Got Pregnant to Quit Smoking: A Randomized Control Trial
Brief Title: A Video-led Smoking Cessation Intervention in Helping Male Smokers Whose Partners Got Pregnant to Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW17-269
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; video; male smoker
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Video+one-sentence smoking cessation advice +general smoking cessation leaflet will be allocated to the participants in the experimental group. The videos which presented the health effects of smoking, especially emphasizing the importance of smoking cessation on the fetal and pregnancy, will be sent in sequence through the smart phone to the participants in the experimental group.
  Interventions: Combination Product: Video+brief smoking cessation+pamphlet
- Conditional control group (Active Comparator): Text-message+one-sentence smoking cessation advice +general smoking cessation leaflet will be allocated to the participants in the experimental group. Text-message contains the same content with videos and will be sent in the same frequency with the videos through the smart phone to the participants in the Conditional control group.
  Interventions: Combination Product: Text-message+brief smoking cessation+pamphlet
- Placebo control group (Placebo Comparator): Participants in the control group will be given a one-sentence smoking cessation advice during the baseline assessment. A leaflet showed the information related to the smoking cessation will be allocated to them at the same time.
  Interventions: Other: brief smoking cessation+pamphlet

INTERVENTIONS:
Combination Product: Video+brief smoking cessation+pamphlet — The videos presented the health effects of smoking, especially emphasizing the importance of smoking cessation on pregnant women, fetuses, and newborns.
  Arms: Experimental group
Combination Product: Text-message+brief smoking cessation+pamphlet — The text -message contains the same content with the videos
  Arms: Conditional control group
Other: brief smoking cessation+pamphlet — The pamphlet showed the general information related to the smoking cessation, the brief smoking cessation only contains a sentence like "You'd better quit smoking."
  Arms: Placebo control group

SUMMARY:
This study aims to use a three arms randomized clinical trial study to evaluate the effectiveness of a video-led intervention in helping male smokers whose partner got pregnant in Mainland China to quit smoking.

DETAILED DESCRIPTION:
With a globally growing number of smokers, up to about half of men and one tenth of women are becoming smokers and relatively few stopping, especially in Mainland China.

It has been proved that tobacco is responsible for even more deaths and diseases. Smokers have two to three times mortality in middle age among otherwise similar persons who had never smoked. According to the literature review, smoking has been confirmed to be an important risk factor to most chronic diseases and cancer.

For the male smokers at their reproductive ages, who is preparing to have a baby, smoking may negatively influence their reproductive capacity. Sufficient studies found that the quantity and duration of smoking, especially the current smoking is positively associated with the risk of erectile dysfunction. Smoking may increase the risk of a higher risk of developing oligospermia, asthenozoospermia and teratozoospermia for man in the reproductive years, which may lead to the inefficiency of fertilization and even give birth to abnormal fetus. Besides, secondhand Smoking (SHS) exposure also have further and longer negative effects on their female partner and their baby born in the future. The non-smoking population is much more sensitive to the nicotine in the passive smoking than smokers. The SHS may increase the risk of respiratory infections, ear problem, immediate adverse effects on cardiovascular system, lung cancer and so on to adults. For the children, the passive smoking make children have a higher chance to get severe asthma, slow lung growth. Hence, children and women live with smokers may have a higher risk of premature death and disease. Besides, newborns whose mothers were exposed to secondhand smoke showed significantly lower scores in the habituation cluster and motor system cluster, as well as the delay of neurobehavioral development regardless of socio-demographic, obstetric and pediatric factors. Conclusively, smoking has direct and indirect negative effect to male smokers in reproductive ages themselves and their family members.

Based on the official statistic figures in 2010, about one third of people in China were current smokers, and the number of young smokers is increasing. While most current smokers (83.9%) report having no intention to quit smoking (WHO, 2011). On average, between 60% and 70% of Chinese men continue to smoke into middle age, which is different with the western countries. Hence, finding out a solution to decrease the married reproductive male smoking rate is extremely crucial.

Overall awareness of the health hazards of tobacco has improved in the last 15 years in China, but is still relatively poor. Even there were several patterns of propaganda and education applied in China, the efficiency is not very satisfactory. Hence, an effective education interventions that delivery the health hazards of tobacco to male smokers and secondhand smoking to their wives and baby born in the future should be developed and implemented for reproductive male smokers in China.

Different patterns of interventions, such as counselling, advertising, leaflets and so on have been implemented, however the effect is not so well as we expected. Thus, a more efficient intervention should be developed. As the high usage rate of smart phone, interventions implemented by cellphone can be considered as a new approach. Watching video has been proven to be significantly associated with prevalence abstinence. Video, combining with the advantage of text, image, and tones, will take visual, auditory and reading stimulation to the brain, consequently, enhance the delivery and memory of information for people. Hence video is an efficient intervention medium for smoking cessation.

Given that, a video-led intervention will be applied to help male smokers whose partner got pregnant in Mainland China to quit or reduce the cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* male resident aged 18 or above;
* smoking at least one cigarette per day averagely during the past 1 months and validated by exhaled CO test (≥ 4ppm);
* have a pregnant partner whose embryo had been confirmed to not have any significant deformity;
* able to communicate in Mandarin (including reading Chinese);
* have a smart phone for intervention and follow-up

Exclusion Criteria:

* smokers who meet the above criteria but are currently involved in other smoking cessation programs or the pilot study;
* mentally or physically unfit for communication;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence at the 6-month follow-up | 6-month follow-up
  The biochemically validated smoking abstinence was confirmed by an exhaled carbon monoxide level < 4 parts per million (p.p.m.)

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 6-month follow-up
  Subjects report that they had not smoked within the recent 7 days.
The level of readiness to quit | 6-month follow-up
  The readiness to quit is divided into pre-contemplation stage (attempt to quit more that 30 days later), contemplation stage (attempt to quit within 30 days but more than 7 days), preparation stage (attempt to quit within 7 days), and action stage (quitting)

CONTACTS AND LOCATIONS:
Overall Officials: William Ho Cheung LI, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia W, Li HCW, Cai W, Song P, Zhou X, Lam KWK, Ho LLK, Cheung AT, Luo Y, Zeng C, Ho KY. Effectiveness of a video-based smoking cessation intervention focusing on maternal and child health in promoting quitting among expectant fathers in China: A randomized controlled trial. PLoS Med. 2020 Sep 29;17(9):e1003355. doi: 10.1371/journal.pmed.1003355. eCollection 2020 Sep. PMID 32991589